CLINICAL TRIAL: NCT02435277
Title: An Extension of Protocol NS-0100-01 to Evaluate the Safety and Effect of Various Fixed-Dose Leucine and Metformin Combinations (NS-0100) Versus Standard Metformin Mono-therapy on Glycemic Control in Subjects With Type 2 Diabetes
Brief Title: An Extension Protocol to Evaluate Dose Comparisons of Leucine-Metformin Combinations in Type 2 Diabetic Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NuSirt Biopharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NS-0100-01E
Record Dates: First submitted 2015-04-13; First posted 2015-05-06 (Estimated); Results first posted 2017-12-18 (Actual); Last update posted 2018-01-17 (Actual); Status verified 2017-12

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Metformin; Leucine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Low Metformin (Experimental): 3 capsules BID with each capsule containing 366.7 mg L-Leucine and 41.7 mg of metformin
  Interventions: Drug: Low Metformin
- Mid Metformin (Experimental): 3 capsules BID with each capsule containing 366.7 mg L-Leucine and 83.3 mg of metformin
  Interventions: Drug: Mid Metformin
- High Metformin (Experimental): 3 capsules BID with each capsule containing 366.7 mg L-Leucine and 166.7 mg of metformin
  Interventions: Drug: High Metformin
- Metformin Monotherapy (Active Comparator): 3 Capsules BID each containing 283.3 mg of metformin BID (1,700 mg/Day) at Day 14.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Low Metformin — 1100 mg L Leucine in combination with 125 mg of Metformin BID
  Other Names: Metformin, L-Leucince, Leucine
  Arms: Low Metformin
Drug: Mid Metformin — 1100 mg L Leucine in combination with 250mg Metformin BID
  Other Names: Metformin, Leucine, L-Leucine
  Arms: Mid Metformin
Drug: High Metformin — 1100 mg of L Leucine in combination with 500 mg Metformin BID
  Other Names: Metformin, Leucine, L-Leucine
  Arms: High Metformin
Drug: Metformin — 500 mg Metformin BID until day 14 with dose escalation at day 14 to 850 mg Metformin BID
  Other Names: Metformin, Leucine, L-Leucine
  Arms: Metformin Monotherapy

SUMMARY:
Study NS-0100-01E is an extension of Study NS-01-0100 designed to assess safety and longer term effect (i.e., additional 8 weeks) of various fixed-dose leucine and metformin combinations (NS-0100) versus standard metformin monotherapy on glycemic control in subjects with type 2 diabetes using HbA1c as the primary endpoint.

DETAILED DESCRIPTION:
This is a randomized, 8-week, extension of Study NS-0100-01, to evaluate the effect of various fixed-dose (FDC) combinations of leucine and metformin compared to standard metformin monotherapy on glycemic control.

Subjects meeting all inclusion criteria and no exclusion criteria for the extension study, including completion of the 4-week treatment period of Study NS-0100-01 [Day 28/Visit 7]), will be eligible to enroll into the extension. During participation in the extension, subjects will continue to receive their assigned treatment based upon the randomization that occurred on Day 1 (Visit 4) of Study NS-0100-0. The study will include a total of 3 visits: Visit 1E (Day 28/Visit 7 of Study NS-0100-01), Visit 2E (Day 56/Week 8), and Visit 3E (Day 84/Week 12). Key assessments at Visit 2E and Visit 3E include HbA1c, fasting plasma glucose, and plasma insulin. In addition, 3-hour standardized meal tests will be performed on Day 28 (as part of the Study Termination [Visit 7] procedures of Study NS-0100-01 prior to enrolling into the extension) and at Study Termination for the extension (Visit 3E [Day 84/Week 12]).

ELIGIBILITY:
Inclusion Criteria:

1. Has completed Study NS-0100-01, including all procedures required at Study Termination (Day 28/Visit 7) without major protocol deviations
2. Is male, or female and, if female, meets all of the following criteria:

   * Not breastfeeding
   * Post-menopausal or negative pregnancy test result (human chorionic gonadotropin, beta subunit [β-hCG]) at Screening (Visit 1) (not required for hysterectomized females)
   * If of childbearing potential (including perimenopausal women who have had a menstrual period within one year) and sexually active, must practice and be willing to continue to practice appropriate birth control (defined as a method which results in a low failure rate, i.e., less than 1% per year, when used consistently and correctly, such as double barrier methods [male condom with spermicide, with or without cervical cap or diaphragm], implants, injectables, oral contraceptives [must have been using for at least the last 3 months], some intrauterine contraceptive devices, tubal ligation, or a vasectomized partner) during the entire duration of the study.
3. Is able to read, understand, and sign the informed consent forms (ICF) and if applicable, an authorization to use and disclose protected health information form (consistent with health insurance portability and accountability act of 1996 [HIPAA] legislation), communicate with the investigator, and understand and comply with protocol requirements.

Exclusion Criteria:

Subjects who meet any of the following criteria will be excluded from the study.

1. Is undesirable as a study participant as judged by the investigator (e.g., exhibited poor compliance during Study NS-0100-01)
2. Is expected to require treatment, or if currently on a stable dose, changes to their regimen of the following medications:

   * Lipid-lowering agents
   * Anti-hypertensive medications
   * Thyroid replacement therapy
   * Non-steroidal anti-inflammatory agents
3. Is expected to require or undergo treatment with any of the following medications:

   * Antidiabetes medications (with the exception of study medication [i.e., metformin])
   * Oral or parenteral steroids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-10; Primary Completion 2015-09 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Orville Kolterman, MD, Study Chair — Pharmapace
Locations (9):
- United States (9):
  - Catalina Research Institute, Chino, California
  - Palm Beach Research, Palm Beach, Florida
  - Meridien Research, Tampa, Florida
  - River Birch Research Alliance, Blue Ridge, Georgia
  - Meridian Research, Savannah, Georgia
  - Streling Research Group, Cincinnati, Ohio
  - Medical Research South, Charleston, South Carolina
  - Meharry Medical College, Nashville, Tennessee
  - Vanderbilt University Medical Center, Diabetes, Endocrinology, and Metabolism, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study NS-0100-01E was a randomized, double-blind 8-week extension of Study NS-0100-01 to evaluate the effect of various fixed-dose combinations of leucine and metformin compared to standard metformin monotherapy on glycemic control.
Pre-assignment Details: Subjects meeting all inclusion criteria and no exclusion criteria for the NS-001-01-E, including completion of the 4-week treatment period of Study NS-0100-01 (Day 28/Visit 7), were eligible to enroll into the NS-001-01-E.
Groups:
- FDC 125: Leucine 1100mg +Metformin 125mg
- FDC 250: Leucine 1100mg +Metformin 250mg
- FDC 500: Leucine 1100mg +Metformin 500mg
- Control: 850mg Metformin
Period: Overall Study
Arm/Group | FDC 125 | FDC 250 | FDC 500 | Control
Started | 12 | 16 | 11 | 11
Completed | 10 | 15 | 11 | 11
Not Completed | 2 | 1 | 0 | 0
Not completed — Adverse Event | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Study NS-0100-01E was the extension of Study NS-01-0100 designed to assess safety and longer term effect (ie, additional 8 weeks) of various fixed-dose leucine and metformin combinations (NS-0100) versus standard metformin monotherapy on glycemic control in subjects with type 2 diabetes.
Groups:
- Total: Total of all reporting groups
Arm/Group | FDC 125 | FDC 250 | FDC 500 | Control | Total
Number analyzed (Participants) | 12 | 16 | 11 | 11 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 13 | 8 | 9 | 40
  >=65 years | 2 | 3 | 3 | 2 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.8 (10.81) | 56.1 (8.24) | 59.8 (9.01) | 60.5 (8.77) | 56.9 (9.52)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 6 | 7 | 29
  Male | 4 | 8 | 5 | 4 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 8 | 2 | 4 | 19
  Not Hispanic or Latino | 7 | 8 | 9 | 7 | 31
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 5 | 4 | 13
  White | 10 | 13 | 6 | 7 | 36
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kg] | 93.343 (19.0179) | 91.314 (18.7664) | 87.497 (21.2259) | 90.500 (18.4163) | 90.782 (18.8230)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: (kg/m^2] | 33.298 (4.4952) | 31.647 (6.3242) | 28.627 (4.5195) | 32.677 (5.3808) | 31.606 (5.4597)
Fasting Plasma Glucose [Mean (Standard Deviation); unit: mg/dL] | 173.5 (31.13) | 150.5 (26.78) | 179.2 (36.04) | 177.1 (53.67) | 168.2 (38.00)
Haemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: %] | 7.56 (0.644) | 7.83 (0.769) | 7.84 (0.545) | 7.92 (0.645) | 7.79 (0.661)
Previous Metformin experience [Count of Participants; unit: Participants]
  No Previous Experience | 2 | 1 | 3 | 2 | 8
  Prior taken metformin: No Abdominal side effects | 9 | 11 | 7 | 8 | 35
  Prior taken metformin: Had abdominal side effects | 1 | 4 | 1 | 1 | 7

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c Levels in Patient Receiving the Various Doses of Leucine and Metformin Combinations
Description: Change in HbA1c from Baseline (Day 1/Visit 1) of Study NS-0100-01 to Week 12 (Day 84/Visit 3E) in subjects receiving various fixed-dose combinations of leucine and metformin compared to standard metformin monotherapy.
Time Frame: Baseline and 12 weeks
Population: Mixed Model Inferential Statistical Analysis of HbA1c change from day 1-day 84 Evaluable Population (n=43)
Measure: Mean (Standard Deviation); unit: percent HbA1c
Arm/Group | FDC 125 | FDC 250 | FDC 500 | Control
Number analyzed (Participants) | 10 | 12 | 11 | 10
percent HbA1c | 0.10 (0.756) | -0.12 (0.987) | -0.05 (0.807) | -0.83 (0.627)
Statistical Analysis 1: Comparison: FDC 125 vs Control; Mixed Model Inferential Statistical Analysis of HbA1c change from day 1-day 84 Evaluable Population (n=43); Test type: Other; p = 0.0475, ANCOVA — Total daily dose is twice the respective dose, Pairwise Comparison using Control as the Reference Group
Statistical Analysis 2: Comparison: FDC 250 vs Control; Test type: Other; p = 0.0912, ANCOVA
Statistical Analysis 3: Comparison: FDC 500 vs Control; Test type: Other; p = 0.0458, ANCOVA

2. Secondary Outcome: Change in Fasting Plasma Glucose
Description: Change in fasting plasma glucose from Baseline (Day 1/Visit 1) of Study NS-0100-01 to Week 12 (Day 84/Visit 3E). Based on the pre-specified mixed model inferential statistical analysis, there was an apparent dose-dependent relationship for the mean decrease from baseline in fasting plasma glucose for the fixed dose leucine amd metformin combination treatments A, B and C.
Time Frame: Baseline and 12 weeks
Population: Mixed Model Inferential Statistical Analysis of Fasting Plasma Glucose change from day 1-day 84 in Evaluable Population (n=43)
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | FDC 125 | FDC 250 | FDC 500 | Control
Number analyzed (Participants) | 10 | 12 | 11 | 10
mg/dL | -15.8 (22.29) | 11.2 (22.37) | -4.3 (39.91) | -36.3 (45.47)
Statistical Analysis 1: Comparison: FDC 125 vs Control; Mixed Model Inferential Statistical Analysis of Fssting Plasma Glucose change from day 1-day 84 in Evaluable Population (n=43); Test type: Other; p = 0.26, ANCOVA — Total daily dose is twice the respective dose Pairwise Comparison using Treatment D as the Reference Group
Statistical Analysis 2: Comparison: FDC 250 vs Control; Test type: Other; p = 0.0083, ANCOVA
Statistical Analysis 3: Comparison: FDC 500 vs Control; Test type: Other; p = 0.0317, ANCOVA

ADVERSE EVENTS:
Time Frame: 84 days
Description: Treatment-Energent Adverse Event (TEAE) is defined as an adverse event occurring on or after the first dose of randomized study medication, or existing prior to the time of and worsening after the time of the first dose of randomized study medication. Subjects experiencing multiple episodes of a given adverse event are counted once. This was a 84 day study and adverse event reporting was upto day 84.
Arm/Group | FDC 125 | FDC 250 | FDC 500 | Control
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/16 | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/12 | 1/16 | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 2/12 | 2/16 | 2/11 | 1/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FDC 125 (N=12) | FDC 250 (N=16) | FDC 500 (N=11) | Control (N=11)
Chest Pain (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FDC 125 (N=12) | FDC 250 (N=16) | FDC 500 (N=11) | Control (N=11)
Gastric Disorders (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Endocrine (Endocrine disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
musculoskeletal (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Respiratory dsorders (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Cough (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Ecchymosis (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hyperglycemia (Endocrine disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes